CLINICAL TRIAL: NCT01717599
Title: Intramuscular Diclofenac in the Prevention of Post-ERCP Pancreatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 4-2012-0466
Record Dates: First submitted 2012-10-25; First posted 2012-10-30 (Estimated); Last update posted 2021-05-04 (Actual); Status verified 2021-05

CONDITIONS: Post ERCP Pancreatitis
Keywords: Post ERCP pancreatitis; Diclofenac; NSAID
MeSH Terms: interventions — Diclofenac; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diclofenac group (Experimental)
  Interventions: Drug: Diclofenac
- Placebo(normal saline) group (Placebo Comparator)
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Diclofenac — Diclofenac 90mg, 2ml/A, IM(intramuscular) injection immediately after procedure of ERCP
  Arms: Diclofenac group
Drug: normal saline — normal saline 2ml/A, IM(intramuscular) injection immediately after procedure of ERCP
  Arms: Placebo(normal saline) group

SUMMARY:
Pancreatitis is one of the major complications of ERCP. It has been shown that NSAIDs are potent inhibitors of phospholipase A2, activity which is increased in pancreatitis. The only one study with IM diclofenac showed reduction of post-ERCP pancreatitis without SOD (sphincter of Oddi dysfunction) by subgroup analysis in small study population. Therefore the investigators must need large scaled randomized control study including of SOD.

DETAILED DESCRIPTION:
The study described in this report will be approved by the ethics committee of Yonsei University School of Medicine, Seoul, Korea. Between July 2012 and February 2013, 380 patients fulfilled the inclusion criteria, 380 of whom were included in the final analysis. Consecutive patients were recruited for the study who presented to the Yonsei University Medical Center with variable symptom or cause for ERCP older than 20years. Patients were excluded from study participation if they had a contraindication for diclofenac, including patients with recently diagnosed peptic ulcer disease or active/recent gastrointestinal hemorrhage within 4 weeks, renal failure(Cr > 1.4), those who had taken an NSAID during the preceding week(ASA 325 mg daily or less acceptable), those who developed acute pancreatitis during the 2 weeks before ERCP, those with a history of chronic calcific pancreatitis or allergy to aspirin or NSAID, and those who did not agree to participate in the study. Additionally, if state of patients was intrauterine pregnancy or breast feeding mother, they were excluded. Entry to the study was restricted to patients advised to have endoscopic retrograde cholangiography with or without pancreatography for extrahepatic cholestasis and/or impaired liver function tests.

The patients received 90 mg IM diclofenac available in our hospital immediately after ERCP at recovery room. Patients were observed in the recovery room for at least 90 minutes after the procedure. Patients in whom abdominal pain developed during this observation period were admitted to the hospital (or for current inpatients, kept in the hospital). Decisions regarding evaluation of complications after the procedure and in-hospital care were left to the discretion of the endoscopist and clinical-service staff members, who were unaware of study-group assignments.

Patients who were discharged after an uneventful ERCP were contacted by telephone within 5 days to capture delayed occurrence of the primary end point. Patient demographics, risk factors, ERCP procedural elements, and follow-up data were recorded on standardized data-collection forms by an investigator or coordinator who was unaware of study-group assignments. The intramuscular route was selected on the basis of available small sized data suggesting that intramuscular NSAIDs are effective in preventing post-ERCP pancreatitis, perhaps owing to more rapid and complete bioavailability than with oral administration. (1) At the end of each procedure, the researchers recorded the details of the maneuvers performed, including the total time of the procedure, the number of attempts at cannulation, the number of pancreatic duct cannulations, the final diagnosis, and whether a sphincterotomy, a needle-knife papillotomy, or stent placement were performed. We did not use pancreatic duct stenting for prevention of pancreatitis. Patients were sedated with IV midazolam and IV continuous infusion of propofol under monitoring by anesthesiologist during whole time of procedure. Xylocaine spray was used as a local anesthetic. Serum amylase was determined 4 hours after ERCP.

If the 4-hours serum amylase level was < 3 times the upper normal limit and there was no clinical evidence of acute pancreatitis at that time, patients were allowed free oral fluids and a diet. If the 4- hours serum amylase level was > 3 times the upper normal limit and the patient exhibited pain or nausea and vomiting, then the patient was kept fasting and IV crystalloid fluids with opiate analgesics were prescribed. The following 24 hours blood tests were repeated for serum amylase and the patients were interviewed and examined for clinical evidence of acute pancreatitis.

Acute pancreatitis was defined as serum amylase at least three times the upper limit of normal range 24hours after the procedure associated with new or increased upper abdomen or epigastric pain, back pain, and epigastric tenderness and hospitalization or prolongation of existing hospitalization for at least 2 nights. Patients with persistent signs and symptoms of pancreatitis after 48 hours underwent contrast-enhanced computed tomography.

Pancreatitis was graded as mild, moderate, or severe. The severity was determined according to consensus guidelines, with mild post-ERCP pancreatitis resulting in a hospitalization of ≤3 days, moderate post-ERCP pancreatitis resulting in a hospitalization of 4-10 days, and severe post-ERCP pancreatitis resulting in a hospitalization of > 10 days, or leading to the development of pancreatic necrosis or pseudocyst, or requiring percutaneous or surgical intervention.

Sphincter of Oddi dysfunction (SOD) was defined according following Classification. Biliary type I SOD was defined as biliary-type abdominal pain, liver enzyme elevation, and common bile duct dilation > 9mm. Biliary type II SOD was defined as biliary-type abdominal pain and either abnormal liver enzymes or a dilated bile duct. Biliary type III SOD was defined as biliary-type pain without any other objective findings. Pancreatic type I SOD was defined as pancreatic-type pain and a dilated pancreatic duct and elevated pancreatic enzymes, or recurrent acute pancreatitis. Type II pancreatic SOD was defined as pancreatic-type pain and a dilated pancreatic duct or elevated pancreatic enzymes. Type III pancreatic SOD was defined as pancreatic-type pain alone.

The instruments used were cannula, sphincterotome, guidewire, and stone basket (Olympus, Japan).

Adverse events were defined as reported previously. Any cases of post-ERCP pancreatitis, other complications of the procedure, and adverse events that were potentially attributable to the study drug were reported to the local institutional review board and the data and safety monitoring board. These reportable adverse events were gastrointestinal bleeding, perforation, infection, renal failure, allergic reaction, myocardial infarction, cerebrovascular accident, and death.

ELIGIBILITY:
Inclusion Criteria:

Consecutive patients were recruited for the study who presented to the Yonsei University Medical Center with variable symptom or cause for ERCP older than 20 years.

Exclusion Criteria:

Patients were excluded from study participation if:

* they had a contraindication for diclofenac,
* including patients with recently diagnosed peptic ulcer disease or active/recent gastrointestinal hemorrhage within 4 weeks,
* renal failure (Cr > 1.4),
* those who had taken an NSAID during the preceding week (ASA 325 mg daily or less acceptable),
* those who developed acute pancreatitis during the 2 weeks before ERCP,
* those with a history of chronic calcific pancreatitis or allergy to aspirin or NSAID, and
* those who did not agree intramuscular injection. Additionally, if state of patients was intrauterine pregnancy or breast feeding mother, they were excluded. Finally, patients were excluded for study if they had bleeding tendency and contraindication for intramuscular injection.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 343 (Actual)
Dates: Start 2012-08-29 (Actual); Primary Completion 2013-08-28 (Actual); Study Completion 2013-08-28 (Actual)

PRIMARY OUTCOMES:
Incidence of post ERCP pancreatitis | 24hours after the procedure(ERCP)
  Acute pancreatitis was defined as serum amylase at least three times the upper limit of normal range 24hours after the procedure associated with new or increased upper abdomen or epigastric pain, back pain, and epigastric tenderness and hospitalization or prolongation of existing hospitalization for at least 2 nights.

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Gastroenterology, Department of Internal Medicine, Yonsei Institute of Gastroenterology, Yonsei University College of Medicine, Seoul, South Korea

REFERENCES:
- [Derived] Park SW, Chung MJ, Oh TG, Park JY, Bang S, Park SW, Song SY. Intramuscular diclofenac for the prevention of post-ERCP pancreatitis: a randomized trial. Endoscopy. 2015 Jan;47(1):33-9. doi: 10.1055/s-0034-1390743. Epub 2014 Nov 19. PMID 25409167